CLINICAL TRIAL: NCT04395976
Title: Effect of Ayurveda as Prophylaxis for Suspected Covid-19 Patients: Randomised Controlled Trial
Brief Title: Ayurveda as Prophylaxis for Suspected COVID-19 Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical approval was denied
Sponsor: British Ayurvedic Medical Council (Other)
Collaborators: All Party Parliamentary Group - Indian Traditional Sciences (Unknown); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAMC01
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Covid-19
Keywords: Ayurveda
MeSH Terms: conditions — COVID-19 | interventions — Medicine, Ayurvedic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants randomised into the control group receive conventional standard care given by recommended guideline.
- Ayurveda (Experimental): Treatment includes a tailored combination of herbs based on individual constitution (based on Ayurveda) nutritional advice, specific consideration of selected food items, specific lifestyle advice, yoga advice along with standard recommendations.
  Interventions: Other: Ayurveda

INTERVENTIONS:
Other: Ayurveda — The Ayurveda intervention is multimodal and following the principles of Ayurveda as a whole medical system, each participants will be treated with individualised care. From the range of proven Ayurvedic Herbs, combination will be decided based on individual participants, his symptoms and his personality.
  Arms: Ayurveda

SUMMARY:
Despite worldwide efforts to contain, manage and treat Covid-19, the pandemic is continuing to spread. This calls for an urgent clinically-proven prophylaxis and therapeutic strategy. Recent developments on the use of traditional medicines in Covid-19 management has drawn enough attention to start several research studies. Based on the Indian Traditional Medicine, Ayurveda's community initiatives, preliminary studies, and our experiential knowledge on Covid-19 settings, we propose present study to prevent the development of COVID-19 symptoms in people who live or have come contact with an individual diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Person who has come into contact with confirmed COVID-19,
* Willing to take study drug as directed

Exclusion Criteria:

* Confirmed current COVID-19
* Inability to take medications orally
* Inability to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical confirmation of Covid-19 | From date of enrolment to 14 days
  Number of participants with symptomatic, lab-confirmed COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Vishwes Kulkarni, Principal Investigator — University of Warwick; Amarjeet S Bhamra, Study Chair — All Party Parliamentary Group - Indian Traditional Sciences; Neha Sharma, Study Director — British Ayurvedic Medical Council
Locations (1):
- British Ayurvedic Medical Council, London, United Kingdom